CLINICAL TRIAL: NCT03016299
Title: The Histological Effect of Various Microfracture Techniques on Human Chondral & Sub-chondral Tissue - an Ex-Vivo Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0167-16-MMC
Record Dates: First submitted 2016-11-16; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-11

CONDITIONS: Partial or Total Hip Arthroplasty; Ex-vivo Preparat of Femoral Head

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Osteoarthritis hip joint: specimen of head of femur will be used- after total hip arthroplasty (due to Degenerative Osteoarthritis hip joint )
  Interventions: Procedure: microfracture techniques
- Non-Osteoarthritis hip joint: specimen of head of femur will be used- after Hip Hemiarthroplasty -Partial replacment (due to traumatic fracture)
  Interventions: Procedure: microfracture techniques

INTERVENTIONS:
Procedure: microfracture techniques — Drill will be performed in 3 contiguous areas. First Area by Nailing, Second by KW drilling and 3rd area drilled by regular drill obtaining a triangle with the three drilled epicenters.

SUMMARY:
The subchondral bone, formed by the subchondral bone plate and the subarticular spongiosa, plays a key role in supporting the articular cartilage. Marrow stimulation techniques such as subchondral drilling are clinically important treatment options for symptomatic small cartilage defects. However, The heat generated from the metal-bone interface during drilling due to the friction can cause thermal osteonecrosis. , recent clinical evidence suggests that they may induce alterations in the subchondral bone plate such as intralesional osteophytes, which persist and may play a role in the degeneration of the repair tissue.

Little is known about whether they induce deleterious changes in the Human Chondral & Subchondral bone.

The aim of this study was to compare the condral & Sub-chondral Histoligical damage induced by different drilling techniques.

To the best of our knowledge this is the first time to inspect it, In- Situ, on Human tissue.

DETAILED DESCRIPTION:
Chronic articular cartilage defects do not heal spontaneously. However, acute traumatic osteochondral lesions or surgically inflicted lesions extending into subchondral bone, spongialization, abrasion or microfracture by drilling causing the release of pluripotent mesenchymal stem cells from the bone marrow, may heal with repair tissue consisting of fibrous tissue, fibrocartilage or hyaline-like cartilage. There for Marrow stimulation techniques as subchondral drilling or microfractures represent ones of the most frequently used methods for chondral and osteochodral defects repair and considered as standard techniques. [10-12]

It's well know and logical to understand that the high temperature around the drilling hole can lead to thermal injury. [1] Temperatures over 47 C degrees for one minutes are associated thermal osteonecrosis [2,3]. The presence of this necrotic bone may delay healing and predispose to infection.[1] Many studies evaluate the thermal necrosis of the drill into the bone [3-6]. In case of osteochondral lesion, drilling of the injury area is the most common practice in orthopedics surgeries for knee, hip, talus and others. In one study that evaluate the difference between drilling and microfractures and the impact in the cartilage healing revealed distinct differences between microfracture and drilling for acute subchondral bone structure and osteocyte necrosis {4] other study evaluate the healing difference between drilling and burring in rabbits knee, showing degenerative changes in both technique and histology longer lived repair the cartilage with 2 mm drilling[5] The main objective of this study is to evaluate for first time in humans, best to our knowledge, the difference between drilling with KWires compared to drill in terms of thermal osteonecrosis and histo-pathological damage.

Methodes:

The specimens will be achieved from 2 groups of patients. The first group correspond to traumatic subcapital fractures with previous non hip pain complains No osteoarthritis changes in the x-ray. The second group the specimens achieve from hip arthroplasty surgery due to osteoarthritic changes.

The femoral head will be obtain during surgery. Drill will be performed in 3 contiguous areas. First Area by Nailing, Second by KW drilling and 3rd area drilled by regular drill obtaining a triangle with the three drilled epicenters. All will be tested with 2 different diameters - 3.5 mm & 1.75mm. All 3 methods will be checked with and without cooling - by laviation with saline during the drilling/nailing. Temperature measurements using Thermocouples having 1 mm wire diameter will be used for temperature measurement.

Parameters as Drilling speed, Drilling depth and Orientation to line of sress- trabeculae- would be uniform.

Histological aspect:

The specimen will be fixed with adequate amount of buffered 4% formalin for 24 to 48 hours with subsequent gentle decalcification in ethylenediaminetetraacetic acid. Then, the specimen will be cut with a strong knife/ or scalpel into parallel slices 3 to 5 mm thick and washed in running water for 12 hours. And after this, the sections from abnormal areas, including articular surface will be submitted for paraffin embedding.

The histological slides will be stained by hematoxilin-eosin (H&E), PAS, Masson trichrome, and Alcian blue. The lesions (degeneration, hemorrhage, necrosis and others) will be measured by micrometer in the microscope.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 who agreed to participate in the study and signed an informed consent form.
* Patients who went through partial or complete arthroplasty of the hip due to traumatic or degenerative changes - respectively.

Exclusion Criteria:

* The refusal of the patient to use sampling for any reason, including the desire for burying the organ / tissue
* rheumatic - autoimmune diseases that may affect the hip joint (eg: psoriasis, rheumatoid arthritis, stc')
* Any chonic medications usage that might affect bone and cartilage (eg: Bifosfantim, Alendronate, Risedronate, Ibandronate)
* Any suspected pathology of bone: malignancies, infections, Avascular Necrosis etc'

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all Adults who went through partial or complete replacement of the hip in our institute
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
histological damage | withing 48 Hours after specimen fixation
  microscopically assesing the histological damage to Human chondral & Subchondral tissue in 3 common microfractures techniques ( morphological description)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alam K. Exploring thermal anisotropy of cortical bone using temperature measurements in drilling. Biomed Mater Eng. 2016 May 12;27(1):39-48. doi: 10.3233/BME-161566. PMID 27175466
- [Background] Augustin G, Davila S, Udilljak T, Staroveski T, Brezak D, Babic S. Temperature changes during cortical bone drilling with a newly designed step drill and an internally cooled drill. Int Orthop. 2012 Jul;36(7):1449-56. doi: 10.1007/s00264-012-1491-z. PMID 22290154
- [Background] Chen H, Hoemann CD, Sun J, Chevrier A, McKee MD, Shive MS, Hurtig M, Buschmann MD. Depth of subchondral perforation influences the outcome of bone marrow stimulation cartilage repair. J Orthop Res. 2011 Aug;29(8):1178-84. doi: 10.1002/jor.21386. Epub 2011 Feb 24. PMID 21671261
- [Background] Chen H, Sun J, Hoemann CD, Lascau-Coman V, Ouyang W, McKee MD, Shive MS, Buschmann MD. Drilling and microfracture lead to different bone structure and necrosis during bone-marrow stimulation for cartilage repair. J Orthop Res. 2009 Nov;27(11):1432-8. doi: 10.1002/jor.20905. PMID 19402150
- [Background] Eriksson AR, Albrektsson T. Temperature threshold levels for heat-induced bone tissue injury: a vital-microscopic study in the rabbit. J Prosthet Dent. 1983 Jul;50(1):101-7. doi: 10.1016/0022-3913(83)90174-9. No abstract available. PMID 6576145
- [Background] Hayashi K, Kumai T, Higashiyama I, Shinohara Y, Matsuda T, Takakura Y. Repair process after fibrocartilaginous enthesis drilling: histological study in a rabbit model. J Orthop Sci. 2009 Jan;14(1):76-84. doi: 10.1007/s00776-008-1284-9. Epub 2009 Feb 13. PMID 19214692
- [Background] Menche DS, Frenkel SR, Blair B, Watnik NF, Toolan BC, Yaghoubian RS, Pitman MI. A comparison of abrasion burr arthroplasty and subchondral drilling in the treatment of full-thickness cartilage lesions in the rabbit. Arthroscopy. 1996 Jun;12(3):280-6. doi: 10.1016/s0749-8063(96)90059-6. PMID 8783821
- [Background] Mohlhenrich SC, Abouridouane M, Heussen N, Holzle F, Klocke F, Modabber A. Thermal evaluation by infrared measurement of implant site preparation between single and gradual drilling in artificial bone blocks of different densities. Int J Oral Maxillofac Surg. 2016 Nov;45(11):1478-1484. doi: 10.1016/j.ijom.2016.05.020. Epub 2016 Jun 11. PMID 27297835
- [Background] Orth P, Goebel L, Wolfram U, Ong MF, Graber S, Kohn D, Cucchiarini M, Ignatius A, Pape D, Madry H. Effect of subchondral drilling on the microarchitecture of subchondral bone: analysis in a large animal model at 6 months. Am J Sports Med. 2012 Apr;40(4):828-36. doi: 10.1177/0363546511430376. Epub 2012 Jan 5. PMID 22223716
- [Background] Singh G, Jain V, Gupta D, Ghai A. Optimization of process parameters for drilled hole quality characteristics during cortical bone drilling using Taguchi method. J Mech Behav Biomed Mater. 2016 Sep;62:355-365. doi: 10.1016/j.jmbbm.2016.05.015. Epub 2016 May 16. PMID 27254280